CLINICAL TRIAL: NCT03637855
Title: Optical Body Composition and Health Assessment (Shape Up! Adults) Study
Brief Title: Shape Up! Adults Study
Status: Completed | Type: Observational
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Other Study IDs: R01DK109008 (NIH)
Record Dates: First submitted 2018-07-19; First posted 2018-08-20 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Identify the unique associations of body shape to body composition indices in a population that represents the variance of sex, age, BMI, and ethnicity found in the US population.

Describe the precision and accuracy of 3DO scans to monitor change in body composition and metabolic health interventions.

Estimate the level of association of 3DO to common health indicators including metabolic risk factors (glucose, triglycerides, HDL-cholesterol, blood pressure, VAT, WC and strength) by gender, race, age, and BMI.

Investigate holistic, high-resolution descriptors of 3D body shape as direct predictors of body composition and metabolic risk using statistical shape models and Latent Class Analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants will be included in the study if they have a self-reported ability to:

  1. walk one-quarter of a mile and climb 10 steps without difficulty,
  2. perform activities of daily living (ADLs) without difficulty, and
  3. have no life-threatening conditions or diseases that would alter their body composition from what is typical for their age, sex, ethnicity, and BMI.

Exclusion Criteria:

* Participants will be excluded if they have any internal metal artifact (e.g. pacemakers, internal fixation, arthroplasty), amputation, physical impairment or previous fracture that would alter body composition assessment or are pregnant or breastfeeding.
* All premenopausal females will be asked for a spot urine sample for pregnancy test prior to participation.
* Those unwilling to comply with this will not be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit a stratified sample of 720 participants, approximately 360 from each site, using the following equally-weighed stratifications: sex, age (18-40, 40-60, 60-80 years), BMI (less than 25, 25-30, 30 and above) and ethnicity (White, Black, Mexican-American, Asian and Native Hawaiian or Other Pacific Islander).
  Within this sample, we will include up to 36 participants with very low and high BMI by special recruitments from our facilities Anorexia Nervosa (AN) and bariatric surgery clinics. The remainder of the participants will be recruited as a sample of convenience using local advertisements around our facilities.
Sampling Method: Non-Probability Sample
Enrollment: 696 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Fat mass | 1 day
  Measure fat mass and percent fat (arms, legs, trunk, and total) using Dual energy X-ray absorptiometry (DXA) data
Lean mass | 1 day
  Measure lean mass (arms, legs, trunk, and total) using Dual energy X-ray absorptiometry (DXA) data
Bone mass | 1 day
  Measure bone mass (arms, legs, lumbar spine, and total) and Bone Mineral Density (spine and total)
Waist to Hip ratio (WHR) from manual tape measurement | 1 day
  Manual physical anthropometry of waist and hip circumferences
Automatic 3D optical (3DO) scan measurement | 1 day
  Automated 3DO measurements generate the following: 476 girth, length, and volume measurements across the whole body.
HUMAC NORM | 1 day
  Will measure isokinetic strength of knee and back to assess muscle function
Jamar hydraulic hand dynamometer | 1 day
  Will measure grip strength to assess muscle function
Fasting glucose levels | 1 day
  Measure fasting glucose levels
Fasting HbA1c levels | 1 day
  Measure fasting HbA1c levels
Fasting insulin levels | 1 day
  Measure fasting insulin levels
Fasting cholesterol levels | 1 day
  Measure fasting cholesterol levels
Fasting triglycerides levels | 1 day
  Measure fasting triglycerides levels

OTHER OUTCOMES:
Fat loss | 24 weeks
  Measure changes in fat mass during intervention using DXA data.
Changes in lean mass | 24 weeks
  Measure changes in lean mass (arms, legs, trunk, and total) during intervention using DXA data
Changes in WHR | 24 weeks
  Measure changes in WHR during intervention
Changes in automatic 3DO scan measurement | 24 weeks
  Changes of automated 3DO measurements during intervention
changes in HUMAC NORM measurement | 24 weeks
  changes of isokinetic strength of knee and back to assess muscle function
changes in Jamar hydraulic hand dynamometer measurement | 24 weeks
  changes of grip strength to assess muscle function
Bioelectrical impedance analysis (BIA) measurements | 1 day
  measurement of the conductance of water, fat, and muscle by placing electrodes on right and left ankles and index fingertips. The analysis measures the amount of water inside cells and outside cells as the amount of muscle and fat.
Body shape from 2D imaging | 1 day
  Through the use of images from a conventional digital camera estimated body dimension will be obtained
Blood pressure levels | 1 day
  Manually measure blood pressure.
Diet History Questionnaire II | 1 day
  The Diet History questionnaire II estimates a participants nutrition intake by asking the participant a series of questions

CONTACTS AND LOCATIONS:
Overall Officials: John Shepherd, PhD, Principal Investigator — University of Hawaii Cancer Research Center
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

REFERENCES:
- [Derived] Marazzato F, McCarthy C, Field RH, Nguyen H, Nguyen T, Shepherd JA, Tinsley GM, Heymsfield SB. Advances in digital anthropometric body composition assessment: neural network algorithm prediction of appendicular lean mass. Eur J Clin Nutr. 2024 May;78(5):452-454. doi: 10.1038/s41430-023-01396-3. Epub 2023 Dec 23. PMID 38142263
- [Derived] Garber AK, Bennett JP, Wong MC, Tian IY, Maskarinec G, Kennedy SF, McCarthy C, Kelly NN, Liu YE, Machen VI, Heymsfield SB, Shepherd JA. Cross-sectional assessment of body composition and detection of malnutrition risk in participants with low body mass index and eating disorders using 3D optical surface scans. Am J Clin Nutr. 2023 Oct;118(4):812-821. doi: 10.1016/j.ajcnut.2023.08.004. Epub 2023 Aug 19. PMID 37598747
- [Derived] Wong MC, Bennett JP, Quon B, Leong LT, Tian IY, Liu YE, Kelly NN, McCarthy C, Chow D, Pujades S, Garber AK, Maskarinec G, Heymsfield SB, Shepherd JA. Accuracy and Precision of 3-dimensional Optical Imaging for Body Composition by Age, BMI, and Ethnicity. Am J Clin Nutr. 2023 Sep;118(3):657-671. doi: 10.1016/j.ajcnut.2023.07.010. Epub 2023 Jul 19. PMID 37474106
- [Derived] McCarthy C, Tinsley GM, Yang S, Irving BA, Wong MC, Bennett JP, Shepherd JA, Heymsfield SB. Smartphone prediction of skeletal muscle mass: model development and validation in adults. Am J Clin Nutr. 2023 Apr;117(4):794-801. doi: 10.1016/j.ajcnut.2023.02.003. Epub 2023 Feb 8. PMID 36822238
- [Derived] Wong MC, Bennett JP, Leong LT, Tian IY, Liu YE, Kelly NN, McCarthy C, Wong JMW, Ebbeling CB, Ludwig DS, Irving BA, Scott MC, Stampley J, Davis B, Johannsen N, Matthews R, Vincellette C, Garber AK, Maskarinec G, Weiss E, Rood J, Varanoske AN, Pasiakos SM, Heymsfield SB, Shepherd JA. Monitoring body composition change for intervention studies with advancing 3D optical imaging technology in comparison to dual-energy X-ray absorptiometry. Am J Clin Nutr. 2023 Apr;117(4):802-813. doi: 10.1016/j.ajcnut.2023.02.006. Epub 2023 Feb 14. PMID 36796647
- [Derived] Wong MC, McCarthy C, Fearnbach N, Yang S, Shepherd J, Heymsfield SB. Emergence of the obesity epidemic: 6-decade visualization with humanoid avatars. Am J Clin Nutr. 2022 Apr 1;115(4):1189-1193. doi: 10.1093/ajcn/nqac005. PMID 35030235
- [Derived] Panizza CE, Wong MC, Kelly N, Liu YE, Shvetsov YB, Lowe DA, Weiss EJ, Heymsfield SB, Kennedy S, Boushey CJ, Maskarinec G, Shepherd JA. Diet Quality and Visceral Adiposity among a Multiethnic Population of Young, Middle, and Older Aged Adults. Curr Dev Nutr. 2020 May 26;4(6):nzaa090. doi: 10.1093/cdn/nzaa090. eCollection 2020 Jun. PMID 33959689
- [Derived] Lowe DA, Wu N, Rohdin-Bibby L, Moore AH, Kelly N, Liu YE, Philip E, Vittinghoff E, Heymsfield SB, Olgin JE, Shepherd JA, Weiss EJ. Effects of Time-Restricted Eating on Weight Loss and Other Metabolic Parameters in Women and Men With Overweight and Obesity: The TREAT Randomized Clinical Trial. JAMA Intern Med. 2020 Nov 1;180(11):1491-1499. doi: 10.1001/jamainternmed.2020.4153. PMID 32986097
- [Derived] Harty PS, Sieglinger B, Heymsfield SB, Shepherd JA, Bruner D, Stratton MT, Tinsley GM. Novel body fat estimation using machine learning and 3-dimensional optical imaging. Eur J Clin Nutr. 2020 May;74(5):842-845. doi: 10.1038/s41430-020-0603-x. Epub 2020 Mar 16. PMID 32203233
- [Derived] Ng BK, Sommer MJ, Wong MC, Pagano I, Nie Y, Fan B, Kennedy S, Bourgeois B, Kelly N, Liu YE, Hwaung P, Garber AK, Chow D, Vaisse C, Curless B, Heymsfield SB, Shepherd JA. Detailed 3-dimensional body shape features predict body composition, blood metabolites, and functional strength: the Shape Up! studies. Am J Clin Nutr. 2019 Dec 1;110(6):1316-1326. doi: 10.1093/ajcn/nqz218. PMID 31553429